CLINICAL TRIAL: NCT02770404
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability, and Pharmacokinetic Study of Single-Ascending Doses of Intravenous Nafithromycin in Healthy Adult Subjects
Brief Title: A Phase 1 Pharmacokinetic Study of Single-Ascending Doses of Intravenous Nafithromycin in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: W-4873-102 SAD study
Record Dates: First submitted 2016-03-09; First posted 2016-05-12 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — nafithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nafithromycin (Experimental): Subjects in Cohorts 1 through 5 receive active treatments. Subjects in Cohort 6 will receive an IV dose of nafithromycin and a single oral dose of nafithromycin in each crossover period.
  Subjects in each of Cohorts 1, 2, and 3 will receive a single dose of 100, 200, or 400 mg, respectively, of nafithromycin on Day 1
  Interventions: Drug: Nafithromycin
- Placebo (Placebo Comparator): Subjects in Cohorts 1 through 5 will be randomly assigned in an 8:2 allocation to receive active or placebo treatments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nafithromycin — 100, 200, or 400 mg of nafithromycin
  Arms: Nafithromycin
Drug: Placebo — IV matching placebo
  Other Names: Matching IV placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, single-center, placebo-controlled, sequential-cohort study in at least 60 healthy adult male and female subjects. Subjects in Cohorts 1 through 5 will be randomly assigned in an 8:2 allocation to receive active or placebo treatments. Subjects in Cohort 6 will be randomly assigned in a 1:1 allocation to receive an IV dose of nafithromycin and a single oral dose of nafithromycin in each crossover period. Subjects in each of Cohorts 1, 2, and 3 will receive a single dose of 100, 200, or 400 mg, respectively, of nafithromycin or matching placebo on Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 18 and 55 years of age, both inclusive,
* creatinine clearance ≥80 mL/minute (Cockcroft-Gault method).

Exclusion Criteria:

1. Clinically relevant pathology or any other systemic disorder/major surgeries that in the opinion of the investigator would confound the subject's participation and follow-up in the clinical study.
2. Drug or food allergy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-12-25 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve | 72 hours from dosing
Maximum observed plasma concentration (Cmax) | 72 hours from dosing
Time to Cmax (Tmax) | 72 hours from dosing

SECONDARY OUTCOMES:
clinical laboratory- Number of subjects with deranged heamatology parameters test results | 14 days
12-lead safety ECG results | 14 days
Number of subjects reported with any local tolerability at the injection site assessments | 14 days
Number of subjects with any abonormal physical examination findings | 14 days
Total number of reported AEs | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Phase 1 unit : Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States